CLINICAL TRIAL: NCT06323863
Title: Ultra-high Resolution CT: the End of Stapes Prosthesis Measurement Misestimation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: N°4-RCB/EUDRACT
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-11

CONDITIONS: Otosclerosis
Keywords: stapes; titanium; computed tomography
MeSH Terms: conditions — Otosclerosis | interventions — Stapes Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent stapes surgery at our instution: patients with otosclerosis who underwent stapedectomy in our institution
  Interventions: Procedure: stapedectomy; Radiation: ultra high resolution CT

INTERVENTIONS:
Procedure: stapedectomy — stapes removal and replacement by a prosthesis
Radiation: ultra high resolution CT — imaging study

SUMMARY:
Actual CT scanners overestimate stapes piston size, and do not represent a valuable technique for their follow-up, especially in case of complication. Ultra-high resolution has not yet been evaluated in this setting.

DETAILED DESCRIPTION:
Modern temporal bone imaging systems, using 0.5 mm slice thickness, are reputed not yet able to depict the stapes piston position with a sufficient degree of accuracy, as high-resolution CT measurements consistently overestimated intravestibular piston dimensions (width by 44%, length by 6.25%) and vestibular intrusion (by 39%) because of metallic artifacts. . The exact limits of intravestibular depth are also unclear. The "safe" intravestibular prosthesis depth varies widely between studies and has been reported to range from 0.2 to 2.5 mm, so 39% may represent up to 0.9 mm of misestimation. Ultra-high resolution CT (UHR-CT) has improved spatial resolution to 0.12 mm by using ultra-small detector elements (0.25 x 0.25 mm), allowing better visualization of temporal bone structures compared to high-resolution temporal bone CT (HR-CT). However, this technique has not been described for stapes prosthesis measurement.

ELIGIBILITY:
Inclusion Criteria:

- stapes prosthesis Ultra-high resolution CT available

Exclusion Criteria:

no materiovigilance report available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with otosclerosis who underwent stapes replacement by a prosthesis and underwent ultra high resolution CT for follow-up
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
length | february 2020 - novembre 2023
  length of the prosthesis on CT

CONTACTS AND LOCATIONS:
Overall Officials: romain gillet, Principal Investigator — CHRU de Nancy
Locations (1):
- Chu Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No
because CT-scanner are the patient's proprety

REFERENCES:
- [Background] Bozzato A, Struffert T, Hertel V, Iro H, Hornung J. Analysis of the accuracy of high-resolution computed tomography techniques for the measurement of stapes prostheses. Eur Radiol. 2010 Mar;20(3):566-71. doi: 10.1007/s00330-009-1582-4. Epub 2009 Sep 2. PMID 19727746
- [Background] Fang Y, Wang B, Galvin JJ 3rd, Tao D, Deng R, Ou X, Liu Y, Dai P, Sha Y, Zhang T, Chen B. MPR-CT Imaging for Stapes Prosthesis: Accuracy and Clinical Significance. Otol Neurotol. 2016 Apr;37(4):321-3. doi: 10.1097/MAO.0000000000000987. PMID 26927761
- [Background] Gil Mun S, Scheffner E, Muller S, Mittmann P, Rademacher G, Mutze S, Wilms K, Boga E, Bjorn Gehl H, Sudhoff H, Todt I. Stapes piston insertion depth and clinical correlations. Acta Otolaryngol. 2019 Oct;139(10):829-832. doi: 10.1080/00016489.2019.1637019. Epub 2019 Jul 12. PMID 31298596